CLINICAL TRIAL: NCT01146509
Title: An Open-Label, Multicenter, One-Year Extension Of The Evaluation Of The Efficacy And Safety Of Donepezil Hydrochloride (E2020) In Migraine Prophylaxis
Brief Title: An Evaluation Of The Efficacy And Safety Of Donepezil Hydrochloride (E2020) In Migraine Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Margaret Moline, Study Director, Eisai Medical Research Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2020-A001-213
Record Dates: First submitted 2009-04-28; First posted 2010-06-17 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Migraine Headache
Keywords: migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Donepezil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Aricept (donepezil hydrochloride)

INTERVENTIONS:
Drug: Aricept (donepezil hydrochloride) — Donepezil hydrochloride tablet: initial 5 mg/day dose was taken orally, once a day. At Week 4 visit, the dose was increased to 10 mg/day at the discretion of the investigator.
  Other Names: donepezil hydrochloride

SUMMARY:
The purpose of this extension study was to evaluate the safety and efficacy of donepezil hydrochloride after extended use in migraine prophylaxis. Efficacy will continue to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have completed study E2020-A001-211 according to the protocol.
2. Male and female patients between 18-65 years of age. Women of childbearing potential practiced effective contraception (e.g., abstinence, intra-uterine device (IUD) or barrier method plus hormonal method), had a negative urine -hCG at Week 0, and be willing to remain on their current form of contraception for the duration of the study. Pregnant and/or lactating females were to be excluded.
3. Patients of any race who were in generally good health.
4. Patient was willing to participate, and has provided written informed consent prior to being exposed to any study-related procedures.

Exclusion Criteria:

1. Evidence of any clinically significant disorder which was being evaluated medically, and which had not been shown to be stable on medications or other treatment(s) for a period of at least 3 months, including active or uncontrolled tumors, non-trauma related cerebrovascular accidents, gastrointestinal, renal, hepatic, endocrine or pulmonary disease, cardiovascular system disease or known collagen vascular disease (e.g., systemic lupus erythematosus). Hypertension was medication controlled (supine diastolic BP < 95 mmHg). Cardiac disease (angina pectoris, congestive heart failure or arrhythmias) was stable on appropriate medication for 6 months. No elective surgical procedures were allowed during the course of the study.
2. Patients with a recent history (</= 2 years) of or on active treatment for any hematologic/oncologic disorders (other than basal or squamous cell carcinoma of the skin).
3. Patients with a serious central nervous system (CNS) disorder (e.g., neoplasm, infection, demyelinating disease, degenerative neurological disease such as Alzheimer's disease, Parkinson's disease, vascular dementia, or any other progressive CNS disease) or who either evidence focal neurological signs or symptoms by examination or history (e.g., papilledema) or who evidence transient neurological symptoms without an ensuing headache.
4. Any medical or psychiatric (e.g., severe depression, psychosis, bipolar disorder) condition which, in the opinion of the Investigator, made the patient unsuitable for the study.
5. History of chronic alcoholism or drug abuse as defined by DSM-IV criteria or patients who had previously been hospitalized and/or treated for substance abuse within the past one year.
6. History of overuse (> 12 days per four week period on average) of acute headache medications including analgesics, opioids, Non-steroidal anti-inflammatory drugs (NSAIDs), butalbital containing compounds, ergots and triptans within the past one (1) year.
7. Patients who were taking any prior or concomitant medications, as defined in the Protocol (Appendix 16.1.1), during the study.
8. Patients who were unwilling or unable to fulfill the requirements of the study.
9. Patients with known hypersensitivity to piperidine derivatives.
10. Patients who had taken a cholinesterase inhibitor (e.g., donepezil, tacrine, rivastigmine, galantamine, metrifonate) for the acute or prophylactic treatment of migraines in the past (excluding E2020-A001-211) or who were currently taking a cholinesterase inhibitor for any other indication.
11. Patients who had taken any unapproved prior or concomitant medications. In particular, patients were not allowed to take beta-blockers, tricyclic antidepressants, calcium channel blockers, monoamine oxidase inhibitors, valproate, methysergide, cyproheptadine or any other ongoing prophylactic treatment for migraines while participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-01; Primary Completion 2004-04 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety: physical examination, vital signs measurement, clinical laboratory evaluation, 12-lead ECG measurement, adverse event (AE) evaluation. | Every visit up to 52 weeks

SECONDARY OUTCOMES:
Proportion of patients experiencing ≥ 50% reduction in migraine frequency per month ("responders"). | Weeks 4, 16, 28, 40 and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Moline, Study Director — Eisai Inc.
Locations (4):
- United States (4):
  - Diamond Headache Clinical, Chicago, Illinois
  - Clinvest/Headache Care Center, Springfield, Missouri
  - Elkind Headache Center, Mount Vernon, New York
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania